CLINICAL TRIAL: NCT05475912
Title: Effect of Talocrural Joint Thrust Manipulation on Mechanical Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01075 Kashmala
Record Dates: First submitted 2022-07-24; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Mechanical Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A, Conventional Pysical Therapy treatment (Experimental): group A will be given, Electrotherapy Modalities treatment:Hot pack - 20 min,Transcutaneous Electrical Nerve Stimulator - 30 min and will perfome Active Exercises including;Knee to chest exercise,Hamstring stretch, Pelvic bridging,Pelvic tilt, Lumbar rotation stretch exercise.(1set with10 reps of each excercise) Home exercise plan & precautions; Perform above mentioned active exercises, 3 sessions per day (1sets x 10 reps) will also be given to Group A.
  Interventions: Other: Group A, excercises
- Group B, Talocrural joint manipulation and Conventional Physical Therapy treatment (Experimental): group Bwill be given, Talocrural Joint Manipulation with Electrotherapy Modalities treatment:Hot pack - 20 min,Transcutaneous Electrical Nerve Stimulator - 30 min and will perfome Active Exercises including;Knee to chest exercise,Hamstring stretch, Pelvic bridging,Pelvic tilt, Lumbar rotation stretch exercise.(1set with10 reps of each excercise) Home exercise plan & precautions; Perform above mentioned active exercises, 3 sessions per day (1sets x 10 reps) will also be given to Group B.
  Interventions: Other: Group A, excercises

INTERVENTIONS:
Other: Group A, excercises — Each group will receive treatment three times per week for 3 weeks total 7 sessions.
  Other Names: Group B,manipulation

SUMMARY:
Among all disabling musculoskeletal condition, non specific low back pain is most prevalent and universal condition. Its prevalence has increased over years and affects almost all at some phase in their life. Though, there are many causes of low back pain such as, sedentary life style, depression, poor nutritionist diet and so on, yet faulty posture is also one of the noteworthy causes of low back pain which cannot be overlooked. Faulty posture can result from any out of order body component, such as atypical foot biomechanics. Since lower limb is connected in a closed chain, atypical foot biomechanics leads to disruption in the whole chain ascending up to the spine, stressing spine soft tissues, upsetting its normal anatomical position and causing low back pain.

DETAILED DESCRIPTION:
The lower limb is made up of all the structures from feet to pelvic, forming a closed mechanical chain. In this chain if any one segment is out of its neutral position it affects the whole chain. Like, if a foot is out of its alignment can be flattened or highly pronated, it will results in ankle internal rotation i,e. during the early stance phase of gait When the foot pronates, the calcaneus everts while the talus adducts and the plantar flexes. This inferomedial translation of the talus, results in inward rotation of shin and knee. Knee internal rotation, then make femur to rotate medially (internally) and pelvic to tilt anteriorly. This increased tilting of pelvic increases the curvature of the lumbar spine. Excessive curve at lumbar spine places excessive strain on the muscles, tendons and ligaments of the lower back, causing them to inflame and resulting pain. This domino effect, explains how a misalignment in the foot end up negatively effecting the health of one's lower back and a source of non specific low back pain.Though the direct treatment of lumbar region is important for LBP,yet ankle strategy is needed in order to correct the spinal imbalance. This research proceeded with the thought of taking a whole approach i.e. treating the main cause, causing LBP rather than just applying specific approach i.e. giving only symptomatic treatment for pain alleviation. With this approch talocrural/ankle joint is being taken within physical therapy treatment sphere through manipulation technique along with conventional physical therapy protocol for LBP in the current study.

ELIGIBILITY:
Inclusion Criteria:

* Participants falling in this category would be recruited into the study.

  * Willingness of participant.
  * Age group between 21-45 years (both male and female).
  * Localized, Low back pain- Sub acute(6-12 weeks) and chronic low back pain(12 weeks and above)
  * Asymptomatic Ankle- Pronated foot, Flat foot, Healed ankle injuries.
  * Test for inclusion of foot: Feiss line test (Medial Longitudinal Arch Angle), Stress Test for Ankle ligaments (Anterior Drawer Test, Talar Tilt Test, Eversion Stress Test).

Exclusion Criteria:

* Participant failing to fall in this category would be excluded of the study.

  * Any recent injury of spine or lower limb.
  * Any unhealed ankle injuries.
  * Patients with neurological deficit such as paresthesia, numbness and weakness in lower limb.
  * Spondylolysis or any defect or stress fracture in the pars interarticularis of the vertebral arch.
  * Spondylolisthesis or any displacement of vertebra.
  * Spinal fracture or any trauma in spinal column.
  * Spinal tumors (both primary and metastatic tumor).
  * Spinal surgery such as lumbar decompression surgery, lumbar fusion surgery.
  * Artificial disc replacement surgery.
  * Pregnancy.
  * Disc prolapsed such as protrusion, prolapse, extrusion and sequestration.
  * Any spinal curvature defect.
  * Receiving steroid injection within previous 3 months.
  * History of systemic disorder and malignancy.
  * Diagnosed diabetic patients.
  * Diagnosed Osteoporotic patients

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | 7 Day
  Effects of Talo-crural joint Thrust Manipulation along with Conventional Physiotherapy Treatment will be observed on Mechanical Low Back Pain, through visual analogue scale.
  Findings suggested that 100-mm VAS ratings of 0 to 4 mm can be considered no pain; 5 to 44 mm, mild pain; 45 to 74 mm, moderate pain; and 75 to 100 mm, severe pain.
  assesment will be made on baseline, before intervention, on 4th session after intervention and on 7th session after intervention.

SECONDARY OUTCOMES:
Modified oswestry disability index | 7 Day
  Effects of Talo-crural joint Thrust Manipulation along with Conventional Physiotherapy Treatment will be observed on quality of life among mechanical low back pain patients, through modified oswestry disability index.
  ODI is made up of 10 questions. Each question is scored from 0-5 (minimum to maximum)
  Assesment will be made on baseline, before intervention, on 4th session after intervention and on 7th session after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmed Awan, PhD, Principal Investigator — Riphah International University Islamabad
Locations (1):
- Kashmala Saleem, Rawalpindi, Punjab Province, Pakistan